CLINICAL TRIAL: NCT03119181
Title: A Prospective, Multicenter Study to Evaluate Effectiveness and Safety of Tymbion Iontophoresis and Tympanostomy Tube Placement Using the Tula Iontophoresis and Tube Delivery Systems for Adults in an Office Setting
Brief Title: Study to Compare Active Tymbion Iontophoresis to Sham Tymbion Iontophoresis for Anesthesia of the Tympanic Membrane
Acronym: ADEPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tusker Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CPR007003 - Group A
Record Dates: First submitted 2017-04-05; First posted 2017-04-18 (Actual); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Lidocaine; Epinephrine; Myo-Inositol-1-Phosphate Synthase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Active Tymbion Iontophoresis (Experimental): Unilateral treatment with active iontophoresis of Tymbion (2% lidocaine HCl/ 1:100,000 epinephrine) using the Tusker Medical Tula Iontophoresis System.
  Interventions: Combination Product: Device: Iontophoresis System (IPS) with Drug: Tymbion lidocaine/epinephrine solution
- Sham Tymbion Iontophoresis (Sham Comparator): The sham iontophoresis procedure will be identical to the active Tymbion iontophoresis in that Tymbion (2% lidocaine/ 1:100,000 epinephrine solution) will be placed in the external ear canal, however the iontophoresis current delivery (which facilitates penetration of drug into the tympanic membrane tissue) will not be activated.
  Interventions: Drug: Tymbion Lidocaine/epinephrine solution

INTERVENTIONS:
Drug: Tymbion Lidocaine/epinephrine solution — The external ear canal will be filled with Tymbion drug solution
  Other Names: 2% lidocaine HCl/ 1:100,000 epinephrine; Tymbion
  Arms: Sham Tymbion Iontophoresis
Combination Product: Device: Iontophoresis System (IPS) with Drug: Tymbion lidocaine/epinephrine solution — The external ear canal will be filled with Tymbion drug solution. The Iontophoresis System (IPS) will be used to deliver current to the Tymbion solution to facilitate drug penetration into the tympanic membrane (TM) tissue to anesthetize (numb) the TM
  Other Names: Tula Iontophoresis System; 2% lidocaine HCl/1:100,000 epinephrine; Tymbion
  Arms: Active Tymbion Iontophoresis

SUMMARY:
A prospective, multicenter study to determine if active Tymbion iontophoresis is superior to sham Tymbion iontophoresis in providing anesthesia to the tympanic membrane (TM). The study will use the Tula iontophoresis systems for healthy adult volunteers in an office setting, called Group A of Protocol CPR007003.

The protocol CPR007003 also includes a Group B study described in a separate Registration (NCT03197558).

DETAILED DESCRIPTION:
The objective of the study is to determine if active Tymbion iontophoresis is superior to sham Tymbion iontophoresis in providing anesthesia to the tympanic membrane. In addition, safety will be evaluated by review of the occurrence of adverse events.

The iontophoresis system (IPS) will be used to facilitate anesthetic delivery to the tympanic membrane (TM). The lidocaine-based solution used for local anesthesia of the TM is Tymbion (2% lidocaine HCl/ 1:100,000 epinephrine).

Group A will consist of 40 evaluable healthy adult subjects randomized (1:1) to receive unilateral treatment (1 ear) with either active Tymbion iontophoresis or sham Tymbion iontophoresis. The sham iontophoresis procedure will be identical to the active Tymbion iontophoresis, with the exception that the iontophoresis current will not be activated (ie, the same drug solution will be applied to ears in both arms). After the completion of the iontophoresis procedure, the tympanic membrane will be tapped with a dull otologic probe to test the level of anesthesia. The subject will rate the level of pain using the Visual Analogue Scale (VAS) immediately after the tap. Investigators and subjects will be blinded to treatment assignment.

Safety assessments will be done post procedure and at follow as applicable.

ELIGIBILITY:
Key Inclusion/Exclusion Criteria

Inclusion Criteria Group A:

1. Healthy adults, 18-50 years old
2. Subject is able and willing to comply with the protocol and attend all study visits
3. Subject is able and willing to provide informed consent
4. Subjects with air conduction hearing thresholds of 25 dB HL or better at standard frequencies up to 2000 Hz, and 45 dB or better at 4000 Hz.
5. Subject is able to read and understand English

Exclusion Criteria Group A:

1. Pregnant or lactating females.
2. Prior ear iontophoresis procedure
3. Subjects with conductive hearing loss.
4. Subjects with history of sensitivity or allergic reaction to lidocaine HCl, tetracaine, epinephrine, or any hypersensitivity to local anesthetics of the amide type, or any component of the anesthetic drug formulation.
5. Familial history of insensitivity to lidocaine or other local anesthetics of the amide type.
6. Significantly atrophic, retracted, bimeric, monomeric or atelectatic tympanic membrane.
7. Perforated tympanic membrane.
8. Subjects with known history of ear surgery or TM condition that has the potential to affect the sensitivity of the TM
9. Otitis externa.
10. Damaged/denuded skin in the auditory canal.
11. Subjects with electrically sensitive support systems
12. Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane.
13. Evidence of Otitis Media at day of procedure, or within the past three (3) months prior to procedure.
14. Other conditions that would preclude performing the study procedure including ear plug incompatibility.
15. Health conditions that, in the opinion of the investigator, would present undue risk to the subject, based on device/anesthetic drug product label warnings and precautions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Camino ENT, San Jose, California
  - Specialty Physician Associates, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Tymbion Iontophoresis | Sham Tymbion Iontophoresis
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Tymbion Iontophoresis | Sham Tymbion Iontophoresis | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (7.7) | 31.9 (7.4) | 30.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 17 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Subject-reported Visual Analog Scale (VAS) Pain Score Following Tympanic Membrane Tap for Subjects Treated With Active Tymbion Iontophoresis Compared to VAS Score for Subjects Treated With Sham Tymbion Iontophoresis.
Description: The VAS consists of a 100 millimeter (mm) line with a statement at each end representing the extreme limits of pain intensity (where 0 represents "No pain" and 100 represents "The worst imaginable pain"). The subject reports their pain intensity by making a mark along the line and the line is measured to convert the subject response to numeric score (0-100 in millimeters). The data will be summarized as the difference in mean VAS scores between the two treatment groups (active Tymbion iontophoresis compared to sham Tymbion iontophoresis).
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Active Tymbion Iontophoresis | Sham Tymbion Iontophoresis
Number analyzed (Participants) | 19 | 21
millimeters | 4.2 (13.1) | 18.3 (24.1)
Statistical Analysis 1: Comparison: Active Tymbion Iontophoresis vs Sham Tymbion Iontophoresis; one-sided permutation test at 2.5% significance; Test type: Superiority; p = 0.0097, one-sided permutation test

ADVERSE EVENTS:
Time Frame: Procedure through 3 days post-procedure
Arm/Group | Active Tymbion Iontophoresis | Sham Tymbion Iontophoresis
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 1/19 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Tymbion Iontophoresis (N=19) | Sham Tymbion Iontophoresis (N=21)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Healthy volunteer experienced a vasovagal episode which resolved prior to start of iontophoresis procedure. The adverse event was reported as mild in severity, non-serious, possibly related to the procedure and unrelated to the drug or device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must submit communications to Sponsor for review and comment to verify accurate content at least 30 days prior to submitting to any third party. A delay up to 90 days may be requested by Sponsor in order to file patent applications relating to an Invention if applicable. Sponsor and PI agree that any Institution Publication shall only be made after the Multicenter Publication, provided that the Multicenter Publication is submitted within 18 months after conclusion of the study at all sites.

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03119181/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT03119181/SAP_001.pdf